CLINICAL TRIAL: NCT02637037
Title: A Two Part Bioequivalence Study to Compare Two Fixed Dose Combination Tablets of Dapagliflozin/Metformin XR 5/500 mg (Part 1) and 10/1000 mg (Part 2) Manufactured at Two Different Plants in Healthy Subjects Under Fasting and Fed Conditions
Brief Title: A Study to Assess the Bioequivalence of Dapagliflozin/Metformin XR Fixed-dose Combination Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1691C00008
Record Dates: First submitted 2015-12-15; First posted 2015-12-22 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Bioequivalence; Fixed Dose Combination Tablets; Healthy Male and Female Subjects
Keywords: dapagliflozin/metformin XR 5/500 mg; dapagliflozin/metformin XR10/1000 mg; bioequivalence; fixed dose combination tablets; pharmacokinetic; type 2 Diabetes Mellitus (T2DM); safety
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Treatment A (Experimental): Under fed conditions, subjects will receive single doses of dapagliflozin/metformin XR test drug (Mount Vernon) 5/500 mg dose
  Interventions: Drug: dapagliflozin/metformin XR 5/500 mg test drug (Mount Vernon)
- Treatment B (Active Comparator): Under fed conditions, subjects will receive single doses of dapagliflozin/metformin XR reference drug (Humacao) 5/500 mg dose
  Interventions: Drug: dapagliflozin/metformin XR 5/500 mg reference drug (Humacao)
- Treatment C (Experimental): Under fasted conditions, subjects will receive single doses of dapagliflozin/metformin XR test drug (Mount Vernon) 5/500 mg dose
  Interventions: Drug: dapagliflozin/metformin XR 5/500 mg test drug (Mount Vernon)
- Treatment D (Active Comparator): Under fasted conditions, subjects will receive single doses of dapagliflozin/metformin XR reference drug (Humacao) 5/500 mg dose
  Interventions: Drug: dapagliflozin/metformin XR 5/500 mg reference drug (Humacao)
- Treatment E (Experimental): Under fed conditions, subjects will receive single doses of dapagliflozin/metformin XR test drug (Mount Vernon) 10/1000 mg dose
  Interventions: Drug: dapagliflozin/metformin XR 10/1000 mg test drug (Mount Vernon)
- Treatment F (Active Comparator): Under fed conditions, subjects will receive single doses of dapagliflozin/metformin XR reference drug (Humacao) 10/1000 mg dose
  Interventions: Drug: dapagliflozin/metformin XR 10/1000 mg reference drug (Humacao)
- Treatment G (Experimental): Under fasted conditions, subjects will receive single doses of dapagliflozin/metformin XR test drug (Mount Vernon) 10/1000 mg dose
  Interventions: Drug: dapagliflozin/metformin XR 10/1000 mg test drug (Mount Vernon)
- Treatment H (Active Comparator): Under fasted conditions, subjects will receive single doses of dapagliflozin/metformin XR reference drug (Humacao) 10/1000 mg dose
  Interventions: Drug: dapagliflozin/metformin XR 10/1000 mg reference drug (Humacao)

INTERVENTIONS:
Drug: dapagliflozin/metformin XR 5/500 mg test drug (Mount Vernon) — single fixed-combination dose tablets
  Arms: Treatment A; Treatment C
Drug: dapagliflozin/metformin XR 5/500 mg reference drug (Humacao) — single fixed-dose combination tablets
  Arms: Treatment B; Treatment D
Drug: dapagliflozin/metformin XR 10/1000 mg test drug (Mount Vernon) — single fixed-dose combination tablets
  Arms: Treatment E; Treatment G
Drug: dapagliflozin/metformin XR 10/1000 mg reference drug (Humacao) — single fixed-dose combination tablets
  Arms: Treatment F; Treatment H

SUMMARY:
This is a bioequivalence study to compare 2 fixed-dose combination tablets of dapagliflozin/metformin XR manufactured at 2 different plants in healthy subjects under fasting and fed conditions

DETAILED DESCRIPTION:
This is a Phase 1, 2-part, open-label, randomized, 4-period, 4-treatment, crossover study in healthy subjects (males and females of non-childbearing potential)

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures
2. Healthy male and female subjects aged 18 - 55 years with suitable veins for cannulation or repeated venipuncture
3. Females must have a negative serum pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling 1 of the following criteria:

   * Post-menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the post-menopausal range
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive at screening

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product
4. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the investigator
5. Any clinically significant abnormal findings in vital signs, as judged by the investigator
6. Any clinically significant abnormalities on 12-lead ECG as judged by the investigator
7. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) antibody
8. Known or suspected history of drug abuse, as judged by the investigator
9. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose.
10. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening
11. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to dapagliflozin/metformin XR.
12. Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening
13. Positive screen for drugs of abuse, cotinine or alcohol at screening or on each admission to the study center
14. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP
15. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, vitamins and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life
16. Known or suspected history of alcohol abuse or excessive intake of alcohol as judged by the investigator
17. Involvement of any AstraZeneca or study site employee or their close relatives
18. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements
19. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2016-04-07 (Actual); Study Completion 2016-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MDCM, M.Sc, CPI, Principal Investigator — PAREXEL Early Phase Clinical Unit Baltimore
Locations (1):
- Research Site, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at PAREXEL International, Early Phase Clinical Unit Baltimore, United States of America. Subjects were randomized into 4-period, 4-treatment (per study part) crossover (4 sequences containing 4 treatments) in fed and fasted state.
Pre-assignment Details: Sequences 1, 2, 3 and 4 Part 1: ABCD, BADC, ABDC, BACD Part 2: EFGH, FEHG, EFHG, FEGH (A = test, fed; B = reference, fed; C = test, fasted; D = reference, fasted; E = test, fed; F = reference, fed; G = test, fasted; H = reference, fasted) A total of 80 subjects were randomized into the study
Groups:
- Part 1: Sequences 1, 2, 3 and 4- each sequence had 10 subjects; Part 1: ABCD, BADC, ABDC, BACD (A = test, fed; B = reference, fed; C = test, fasted; D = reference, fasted) Part 1: Test: Dapagliflozin/metformin XR mg manufactured at Mount Vernon plant (1 x 5/500 mg); Reference: Dapagliflozin/metformin XR mg manufactured at Humacao plant (1 x 5/500 mg)
- Part 2: Sequences 1, 2, 3 and 4 - each sequence had 10 subjects Part 2: EFGH, FEHG, EFHG, FEGH (E = test, fed; F = reference, fed; G = test, fasted; H = reference, fasted) Part 2: Test: Dapagliflozin/metformin XR manufactured at Mount Vernon plant (1 x 10/1000 mg); Reference: Dapagliflozin/metformin XR manufactured at Humacao plant (1 x 10/1000 mg)
Period: Overall Study
Arm/Group | Part 1 | Part 2
Started | 40 | 40
Completed | 36 | 39
Not Completed | 4 | 1
Not completed — Positive drug screen at admission | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.4 (10.38) | 38.1 (9.71) | 36.5 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 39 | 37 | 76

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration-time Curve [AUC] Under Fasted or Fed State
Description: To evaluate the Bioequivalence for Dapagliflozin and Metformin following administration Dapagliflozin/Metformin XR 5/500 mg and 10/1000 mg Manufactured at Mt. Vernon plant, US, Compared to Humacao plant, Puerto Rico, in the Fasted or Fed state.
Time Frame: Days 1 to 3: pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose for each treatment period
Population: PK Analysis Set: All subjects in the safety analysis set for whom at least one of the primary PK parameters could be calculated for at least one analyte (dapagliflozin or metformin), and who had no major protocol deviations thought to impact on analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Treatment A: Fed - 5/500 mg - Dapagliflozin/metformin XR mg manufactured at Mount Vernon plant
- Treatment B: Fed - 5/500 mg - Dapagliflozin/metformin XR mg manufactured at Humacao plant
- Treatment C: Fasted - 5/500 mg - Dapagliflozin/metformin XR manufactured at Mount Vernon plant
- Treatment D: Fasted - 5/500 mg - Dapagliflozin/metformin XR manufactured at Humacao plant
- Treatment E: Fed - 10/1000 mg - Dapagliflozin/metformin XR manufactured at Mount Vernon plant
- Treatment F: Fed - 10/1000 mg - Dapagliflozin/metformin XR manufactured at Humacao plant
- Treatment G: Fasted - 10/1000 mg - Dapagliflozin/metformin XR manufactured at Mount Vernon plant
- Treatment H: Fasted - 10/1000 mg - Dapagliflozin/metformin XR manufactured at Humacao plant
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F | Treatment G | Treatment H
Number analyzed (Participants) | 40 | 38 | 37 | 36 | 37 | 39 | 39 | 39
h*ng/mL
  Dapagliflozin | 236.3 (21.06) | 248.6 (20.79) | 251.6 (21.20) | 258.2 (18.35) | 471.9 (27.46) | 486.9 (26.47) | 504.4 (27.22) | 516.6 (27.15)
  Metformin: number analyzed (Participants) | 37 | 34 | 31 | 30 | 37 | 38 | 36 | 37
  Metformin | 5484 (24.69) | 5465 (27.87) | 4398 (29.41) | 4460 (29.69) | 8403 (27.90) | 8015 (31.65) | 7727 (30.82) | 7578 (35.76)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Dapagliflozin: Statistical Assessment of Bioequivalence for Dapagliflozin following administration Dapagliflozin/Metformin XR 5/500 mg for Treatment A and B; Test type: Non-Inferiority or Equivalence — If the 90% CIs for both dapagliflozin and metformin geometric mean ratio of AUC is entirely contained within an 80.00% to 125.00% interval, it will be concluded the 2 manufacturing sites are bioequivalent; Ratios of Geometric means = 0.96, 90% CI 2-sided [0.93 to 0.99]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Dapagliflozin: Statistical Assessment of Bioequivalence for Dapagliflozin following administration Dapagliflozin/Metformin XR 5/500 mg for Treatment C and D; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.99, 90% CI 2-sided [0.96 to 1.01]
Statistical Analysis 3: Comparison: Treatment E vs Treatment F; Dapagliflozin: Statistical Assessment of Bioequivalence for Dapagliflozin following administration Dapagliflozin/Metformin XR 10/1000 mg for Treatment E and F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.97, 90% CI 2-sided [0.94 to 1.00]
Statistical Analysis 4: Comparison: Treatment G vs Treatment H; Dapagliflozin: Statistical Assessment of Bioequivalence for Dapagliflozin following administration Dapagliflozin/Metformin XR 10/1000 mg for Treatment G and H; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.98, 90% CI 2-sided [0.95 to 1.00]
Statistical Analysis 5: Comparison: Treatment A vs Treatment B; Metformin: Statistical Assessment of Bioequivalence for Metformin following administration Dapagliflozin/Metformin XR 5/500 mg for Treatment A and B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 1.01, 90% CI 2-sided [0.96 to 1.06]
Statistical Analysis 6: Comparison: Treatment C vs Treatment D; Metformin: Statistical Assessment of Bioequivalence for Metformin following administration Dapagliflozin/Metformin XR 5/500 mg for Treatment C and D; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 1.00, 90% CI 2-sided [0.93 to 1.07]
Statistical Analysis 7: Comparison: Treatment E vs Treatment F; Metformin: Statistical Assessment of Bioequivalence for Metformin following administration Dapagliflozin/Metformin XR 10/1000 mg for Treatment E and F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 1.05, 90% CI 2-sided [0.99 to 1.11]
Statistical Analysis 8: Comparison: Treatment G vs Treatment H; Metformin: Statistical Assessment of Bioequivalence for Metformin following administration Dapagliflozin/Metformin XR 10/1000 mg for Treatment G and H; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 1.03, 90% CI 2-sided [0.96 to 1.10]

2. Primary Outcome: AUC From Time Zero to Time of Last Quantifiable Concentration [AUC (0-t)] Under Fasted or Fed State.
Description: as for outcome 1
Time Frame: Days 1 to 3: pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose for each treatment period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F | Treatment G | Treatment H
Number analyzed (Participants) | 40 | 38 | 37 | 36 | 39 | 40 | 39 | 39
h*ng/mL
  Dapagliflozin | 228.1 (20.43) | 239.1 (21.10) | 243.4 (20.93) | 248.8 (17.92) | 454.7 (27.15) | 472.1 (26.72) | 490.9 (27.30) | 505.1 (26.80)
  Metformin | 5307 (26.54) | 5205 (28.59) | 4211 (28.71) | 4212 (27.22) | 8040 (27.82) | 7798 (32.77) | 7456 (30.57) | 7401 (34.75)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.96, 90% CI 2-sided [0.94 to 0.99]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.99, 90% CI 2-sided [0.97 to 1.02]
Statistical Analysis 3: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.96, 90% CI 2-sided [0.93 to 0.98]
Statistical Analysis 4: Comparison: Treatment G vs Treatment H; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.97, 90% CI 2-sided [0.95 to 1.00]
Statistical Analysis 5: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 1.02, 90% CI 2-sided [0.97 to 1.08]
Statistical Analysis 6: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 6]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 1.01, 90% CI 2-sided [0.95 to 1.06]
Statistical Analysis 7: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 1, analysis 7]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of geometric means = 1.03, 90% CI 2-sided [0.97 to 1.09]
Statistical Analysis 8: Comparison: Treatment G vs Treatment H; [analysis description as in outcome 1, analysis 8]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 1.01, 90% CI 2-sided [0.95 to 1.07]

3. Primary Outcome: Observed Maximum Plasma Concentration [Cmax] Under Fasted or Fed State
Description: as for outcome 1
Time Frame: Days 1 to 3: pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose for each treatment period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F | Treatment G | Treatment H
Number analyzed (Participants) | 40 | 38 | 37 | 36 | 39 | 40 | 39 | 39
ng/mL
  Dapagliflozin | 39.69 (26.42) | 41.33 (18.49) | 65.28 (25.49) | 67.41 (24.95) | 87.48 (30.14) | 90.14 (32.09) | 125.6 (30.77) | 132.7 (28.31)
  Metformin | 510.2 (22.23) | 503.4 (22.16) | 563.2 (30.27) | 573.9 (28.55) | 982.6 (28.11) | 975.5 (27.89) | 1016 (35.36) | 998.5 (36.05)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.98, 90% CI 2-sided [0.93 to 1.03]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.97, 90% CI 2-sided [0.90 to 1.06]
Statistical Analysis 3: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.97, 90% CI 2-sided [0.89 to 1.05]
Statistical Analysis 4: Comparison: Treatment G vs Treatment H; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.95, 90% CI 2-sided [0.87 to 1.03]
Statistical Analysis 5: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 1.01, 90% CI 2-sided [0.96 to 1.07]
Statistical Analysis 6: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 6]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 0.98, 90% CI 2-sided [0.92 to 1.04]
Statistical Analysis 7: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 1, analysis 7]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of geometric means = 1.00, 90% CI 2-sided [0.95 to 1.06]
Statistical Analysis 8: Comparison: Treatment G vs Treatment H; [analysis description as in outcome 1, analysis 8]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratios of Geometric means = 1.02, 90% CI 2-sided [0.94 to 1.10]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (t Max)
Description: To characterize and compare the pharmacokinetic profiles of dapagliflozin and metformin when administered as the 2 fixed-dose combination formulations and in the fed and fasted states.
Time Frame: Days 1 to 3: pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose for each treatment period
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F | Treatment G | Treatment H
Number analyzed (Participants) | 40 | 38 | 37 | 36 | 39 | 40 | 39 | 39
Hour
  Dapagliflozin | 2.50 [1.00 to 4.00] | 3.00 [1.00 to 4.00] | 1.00 [0.50 to 2.98] | 1.00 [0.48 to 2.92] | 2.00 [0.98 to 4.00] | 2.00 [0.98 to 4.00] | 1.00 [0.50 to 1.98] | 1.00 [0.48 to 3.00]
  Metformin | 6.00 [4.00 to 11.95] | 6.00 [3.98 to 12.03] | 4.00 [2.00 to 6.00] | 4.00 [2.00 to 6.03] | 4.00 [3.98 to 7.98] | 4.00 [3.98 to 6.02] | 4.00 [1.00 to 6.00] | 4.00 [1.98 to 6.00]

5. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve [t½λz]
Description: as for outcome 4
Time Frame: Days 1 to 3: pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose for each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F | Treatment G | Treatment H
Number analyzed (Participants) | 40 | 38 | 37 | 36 | 39 | 40 | 39 | 39
Hour (h)
  Dapagliflozin: number analyzed (Participants) | 40 | 38 | 37 | 36 | 39 | 39 | 38 | 39
  Dapagliflozin | 14.01 (6.747) | 14.65 (7.245) | 13.73 (6.203) | 16.55 (8.260) | 14.88 (6.272) | 14.42 (5.778) | 14.72 (5.641) | 15.11 (5.998)
  Metformin: number analyzed (Participants) | 34 | 32 | 29 | 26 | 31 | 33 | 31 | 36
  Metformin | 13.48 (7.873) | 12.87 (6.587) | 11.91 (7.351) | 13.52 (8.760) | 14.18 (7.718) | 13.74 (6.984) | 14.38 (8.241) | 15.94 (9.671)

6. Secondary Outcome: Apparent Total Body Clearance After Extravascular Administration Estimated as Dose Divided by AUC [CL/F]
Description: as for outcome 4
Time Frame: Days 1 to 3: pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose for each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F | Treatment G | Treatment H
Number analyzed (Participants) | 40 | 38 | 37 | 36 | 39 | 40 | 39 | 39
L/h
  Dapagliflozin: number analyzed (Participants) | 40 | 38 | 37 | 36 | 37 | 39 | 39 | 39
  Dapagliflozin | 421.3 (194.2) | 424.4 (217.3) | 412.7 (220.5) | 454.6 (202.6) | 476.5 (224) | 433.3 (196.1) | 441.7 (191.7) | 421.4 (163.1)
  Metformin: number analyzed (Participants) | 40 | 34 | 31 | 30 | 39 | 40 | 36 | 37
  Metformin | 2030 (1407) | 2133 (1891) | 2104 (1309) | 2803 (2066) | 3357 (2549) | 3324 (2713) | 3635 (2648) | 3212 (2079)

7. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration [Vz/F]
Description: as for outcome 4
Time Frame: Days 1 to 3: pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose for each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F | Treatment G | Treatment H
Number analyzed (Participants) | 40 | 38 | 37 | 36 | 39 | 40 | 39 | 39
L
  Dapagliflozin: number analyzed (Participants) | 40 | 38 | 37 | 36 | 37 | 39 | 39 | 39
  Dapagliflozin | 21.62 (4.617) | 20.55 (4.506) | 20.32 (4.503) | 19.68 (3.650) | 21.93 (5.747) | 21.22 (5.585) | 20.49 (5.138) | 20.00 (4.974)
  Metformin: number analyzed (Participants) | 40 | 34 | 31 | 30 | 39 | 38 | 36 | 37
  Metformin | 93.78 (22.71) | 94.89 (26.81) | 118.1 (32.16) | 116.9 (36.62) | 123.5 (34.68) | 130.5 (39.23) | 134.9 (37.59) | 140 (50.70)

ADVERSE EVENTS:
Time Frame: From screening until 72 hours postdose for each treatment period (ie. visit 1 to visit 6).
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F | Treatment G | Treatment H
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38 | 0/37 | 0/36 | 0/39 | 0/40 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 2/40 | 5/38 | 1/37 | 2/36 | 2/39 | 4/40 | 4/39 | 3/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=40) | Treatment B (N=38) | Treatment C (N=37) | Treatment D (N=36) | Treatment E (N=39) | Treatment F (N=40) | Treatment G (N=39) | Treatment H (N=39)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.